CLINICAL TRIAL: NCT06444074
Title: The PACT (Patient Activation Through Conversations) Study - A Cluster Randomised Trial of a Health Coach-led Patient Activation Program in Type 2 Diabetes.
Brief Title: The PACT (Patient Activation Through Conversations) Study
Acronym: PACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00667
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Health Coaching; Endocrinology; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study design is a pragmatic cluster randomised controlled trial. Each cluster consists of a Teamlet in a National Health Group Polyclinic (NHGP), consisting of a regular group of Family Physicians, a Care Manager, and a Care Coordinator, that provide chronic care for a regular group of about 5000 patients.
  Teamlets in each polyclinic will be randomised to either the PACT Program condition or Usual Care condition. Patients who belong to Teamlets that are randomised to the PACT Program condition will be recruited for participation in the PACT Program, and patients who belong to Teamlets that are randomised to the Usual Care condition will be recruited and provided with routine care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT Arm (Experimental): Participants in the intervention arm will undergo the PACT Program, which is a 3-month long health coaching program.
  Interventions: Behavioral: Patient Activation through Conversations (PACT) Program
- Usual Care (Placebo Comparator): Patients in the Usual Care Arm will undergo routine follow-up for their Diabetes Mellitus. In NHGP, this involves Teamlet care, where patients are taken care of by a team comprising of Family Physicians, a Care Manager (a nurse trained in chronic disease management), and a Care Coordinator, and are seen typically every three to six months for monitoring of their diabetic control.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Patient Activation through Conversations (PACT) Program — Participants in the intervention arm will undergo a 3-month long health coaching program where a care coach will review a participant's health parameters and current self-care behaviours, identify health motivators and set goals for improving their diabetes, as well as fortnightly support through text or phone call.
  Arms: PACT Arm
Behavioral: Usual Care — Routine Chronic Disease care
  Arms: Usual Care

SUMMARY:
The PACT Study is a cluster randomised trial of a health coach-led patient activation program in type 2 diabetes. The goal of this clinical trial is to evaluate the effectiveness of a health coaching intervention (PACT program) led by Care Coaches (trained lay persons), in adult participants with sub-optimally controlled Diabetes Mellitus, as compared to participants undergoing routine care for diabetes (Usual Care).

The primary outcome of interest is change in Glycated Haemoglobin (HbA1c) levels over 3 months, 6 months and 12 months. Secondary outcomes include changes in blood pressure, low-density lipoprotein-cholesterol (LDL-C) levels, body mass index (BMI), self-reported diabetes self-care behaviours, self-efficacy, health-related quality of life, and diabetes-related distress, over 3, 6 and 12 months.

Participants in the Intervention arm will undergo the PACT Program, which is a 3-month long health coaching program led by a care coach. Participants review their motivators, health parameters, self-care behaviours, and set goals for improving their diabetes using a PACT report. Subsequently, they will receive fortnightly motivational and problem solving support via telephone or WhatsApp messaging over a 3-month duration, and will return to routine care after 3 months. Participants in the Usual Care arm will have routine care of their diabetes treatment.

DETAILED DESCRIPTION:
Study Methodology

This is a cluster randomised controlled trial comparing the PACT program to Usual Care. Each cluster consists of a Teamlet in a NHG Polyclinic, consisting of a regular group of Family Physicians, a Care Manager, and a Care Coordinator, that provide chronic care for a regular group of about 5000 patients.

Study Population

The study population will include patients with suboptimal control of diabetes (HbA1c >8%) between the ages of 21 to 64. Patients with a suboptimal control of diabetes frequently require a combination of both pharmacological and lifestyle measures for improvement of their glycaemic levels.

The inclusion criteria include the following:

* Individuals with a diagnosis of Type 2 Diabetes Mellitus who are enrolled in Teamlets in NHGP
* Age between 21 to 64 years old
* HbA1c level of more than 8% in the last 6 months

The exclusion criteria includes the following:

* History of acute coronary syndrome in the past 3 months
* History of stroke or transient ischaemic attacks in the past 3 months
* History of end stage organ failure (liver cirrhosis, cardiac failure, latest eGFR <30 mL/min/1.73m2 in the last 6 months)
* Cancer requiring treatment in the past 5 years.
* Active psychiatrist follow up
* Social issues that are significant enough for follow-up or referral with a medical social worker within the last 12 months
* Women who are pregnant or breastfeeding
* Patients who are enrolled in other current diabetes-related interventional studies
* Inability to provide written consent for the study protocol and able to commit to the study duration.

These patients are excluded as they may have conditions that could be of a higher priority for management as compared to Diabetes Mellitus, and may not be able to provide informed consent or participate actively in shared decision making.

Summary of Study Design

The unit of randomisation will be each cluster, as represented by a single Teamlet. Randomisation will be carried out on all Teamlets that are involved in this research study from NHG Polyclinics. The study team aims to involve two to three polyclinics that includes six Teamlets in each polyclinic. A total of 12 to 18 Teamlets will hence be involved, subject to resource and recruitment considerations.

Teamlets in each polyclinic will be randomised to either the PACT Program condition or Usual Care condition. Patients who belong to Teamlets that are randomised to the PACT Program condition will be recruited for participation in the PACT Program, and patients who belong to Teamlets that are randomised to the Usual Care condition will be recruited and provided with routine care. Due to the nature of the PACT intervention, blinding of the Teamlet members (Doctor, Care Manager, Care Coach) and patients will not be feasible. The data analyst will be blinded to the group allocation.

The PACT Program intervention will last 3 months. Four participant assessments will be conducted, and this will take place at baseline and at the 3-month, 6-month, and the 12-month mark.

Recruitment of participants will take place over 12 months and follow-up of participants will be carried out over 24 months. Further analysis will be undertaken for 12 months, so the total length of the study will be 4 years and 0 months.

PACT program procedures The PACT program lasts 3 months and is a health coaching program for people with type 2 diabetes.

Patients have an in-person visit with a Care Coach at the baseline visit, where review of their metabolic parameters, self-care behaviors and health motivators is carried out, supported by use of a PACT form. This is followed by goal setting.

The PACT form consists of:

1. Results of patients' latest clinical readings are shared with the patient
2. Patient fills in their key motivators for managing their diabetes well
3. Patient fills in a survey that assesses their own self-care behaviors (diet, exercise, medication adherence), diabetes distress
4. Goal setting with the care coach to set SMART (specific, measurable, achievable, relevant and time-sensitive) goals

The Care Coach has been trained to apply a bio-psychosocial approach, motivational interviewing skills and provide diabetes care support. The discussion will take approximately 15 to 30 minutes.

Supportive follow-up is provided over the following 3 months. The Care Coach will support patients in reviewing their goals, assist in problem solving, and provide motivational support. Follow-up will be conducted 2 weekly via telephone calls and/or WhatsApp messages, according to the patient's preference. Care coaches will minimally send patients a whatsapp message or conduct a phone call, however, we acknowledge that some patients may not reply or pick up the phone. This will take approximately 10 to 20 minutes each time. After 3 months, the patients will be reverted back to routine clinical care.

Outcome Assessments

Patient outcomes will be assessed at baseline (12 months before study period), and at regular intervals over 24 months for clinical data. Patient reported outcomes will be assessed at 3, 6, and 12 months.

1. Clinical Outcomes

   * Clinical outcomes will be extracted from the NHGP Business Intelligence database, from routinely collected data.
   * The outcomes that will be assessed include:

     * Clinical outcomes at baseline and follow-up: HbA1c, systolic and diastolic blood pressure, body mass index, Total cholesterol, HDL-cholesterol, LDL-cholesterol, and Triglyceride levels, serum creatinine level, estimated glomerular filtration rate, urine albumin-creatinine ratio, and the urine protein-creatinine ratio
     * At baseline: Presence of co-morbidities, which include hypertension, hyperlipidaemia, ischaemic heart disease, stroke, peripheral vascular disease, previous lower limb amputations, chronic kidney disease, diabetic neuropathy, and diabetic retinopathy
   * Patients usually make clinic visits every 3 to 6 months. Clinical outcomes data will be obtained for baseline and over a period of 24 months.
2. Patient reported outcomes

   * Patient reported outcomes will be assessed using a questionnaire at baseline, at the 3-month mark, 6-month mark, and at the 12-month mark.
   * The questionnaire will be self-administered with interviewer assistance on patient request.
   * The baseline and follow-up questionnaires include the following measures:

     * Sociodemographic information - Only in baseline questionnaire
     * Self-care behaviours, measured with the Summary of Diabetes Self-Care Activities scale (SDSCA)
     * Diabetes-related distress, measured with the 2-item Diabetes Distress Scale (DDS-2)
     * Diabetes empowerment, measured with the short form of the Diabetes Empowerment Scale (DES-SF)
     * Health-related quality of life, measured with the EQ-5D-5L
     * Patient satisfaction, as measured by 5 questions from the Patient Satisfaction Questionnaire-III- Only in the PACT 3-month questionnaire.
3. Referral to community exercise programs. As part of comprehensive lifestyle management, the patients may be directed to community exercise programs, such as those run by SportSG. Attendance to such programs will be recorded via patient-reported information in the 3-month, 6-month, and 12-month questionnaires.
4. Adverse events Improvements in self-care behaviors (diet and physical activity) may be associated with hypoglycaemic symptoms. Monitoring for serious hypoglycaemic episodes requiring emergency department visit and/or admissions to hospital will be recorded via patient-reported information the 3-month, 6-month, and 12-month questionnaires.
5. Drugs Prescribed Drugs could affect clinical outcomes such as HbA1c. Information such as drug prescribed, dosage, and cost of medications will be extracted from NHGP Business Intelligence database.
6. Resources and Cost

Costs and resource utilisation will be analysed, including:

* Health-service utilisation costs including Medical (Doctor), Nursing (Care Manager), Allied Health (Dietician, Psychologist, Medical Social Worker) consultation sessions
* Training and utilisation costs for the Care Coaches, including the number of Telephone/WhatsApp follow-up calls by the Care Coaches
* Laboratory tests
* Medication costs

Sample Size and Statistical Methods

Estimation of Sample Size A minimal clinically important difference of 0.4% in HbA1c is expected between participants of the PACT program compared with Usual Care. In estimating the sample size, a standard deviation of 1.2% was used, as estimated from a local study. We aim to recruit between 12 to 18 Teamlets in the study. If 12 Teamlets are recruited (6 Teamlets are randomised to PACT and 6 to the control group), 34 subjects are required for each Teamlet (total 204 participants in the PACT program and 204 participants in Usual Care), at 80% power with one-sided alpha at 5%, and setting the intracluster correlation coefficient at 0.01 with an assumed drop-out rate of 20%. If 18 Teamlets are recruited (9 randomised to PACT and 9 to the control group), 24 subjects are required for each Teamlet (216 participants in the PACT program and 216 participants in Usual Care), at 80% power with one-sided alpha at 5%, and setting the intracluster correlation coefficient at 0.01 with an assumed drop-out rate of 20%. Sample size calculations were conducted using SampSizeV2.

Statistical and Analytical Plans

1. Clinical Outcomes evaluation Categorical data will be summarized as counts (percentage), while continuous data will be summarized as mean (standard deviation) if they are normally distributed or median (interquartile range) if they are skewed. Baseline characteristics will be compared between participants in the PACT program and Usual care. Differences in the outcomes of interest (clinical and patient-reported) at different data points will be compared between participants in the PACT program and Usual Care. As this is a cluster-randomised trial, a mixed model will be used to evaluate the longitudinal difference-in-difference outcomes between the PACT program and Usual Care, incorporating Teamlets as the random effect. Relevant baseline covariates will be included in the model to account for potential confounding factors.
2. Resource and cost evaluation This study will analyse the cost-effectiveness and resource utilisation of the PACT program. The potential economic impact of new program implementation will be studied by estimating the incremental cost effectiveness ratio (ICER) between PACT and Usual Care (incremental direct medical cost per unit improvement in clinical outcome).

Effectiveness outcomes may include differences between PACT and controls in terms of HbA1c, DM-related complications, DM-related deaths, or quality-adjusted life years (QALYs).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of Type 2 Diabetes Mellitus who are enrolled in Teamlets in NHGP
* Age between 21 to 64 years old
* HbA1c level of more than 8% in the last 6 months

Exclusion Criteria:

* History of acute coronary syndrome in the past 3 months
* History of stroke or transient ischaemic attacks in the past 3 months
* History of end stage organ failure (liver cirrhosis, cardiac failure, latest eGFR <30 mL/min/1.73m2 in the last 6 months)
* Cancer requiring treatment in the past 5 years.
* Active psychiatrist follow up
* Social issues that are significant enough for follow-up or referral with a medical social worker within the last 12 months
* Women who are pregnant or breastfeeding
* Patients who are enrolled in other current diabetes-related interventional studies
* Inability to provide written consent for the study protocol and able to commit to the study duration.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 432 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2028-04-22 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 24 Months
  Glycated Hemoglobin

SECONDARY OUTCOMES:
Blood Pressure | 24 months
  Systolic and Diastolic Blood Pressure
BMI | 24 months
  Body Mass Index
LDL-C | 24 months
  Low density Lipoprotein cholesterol
eGFR | 24 months
  Estimated glomerular filtration rate
uACR | 24 months
  Urine Albumin:Creatinine Ratio
uPCR | 24 months
  Urine Protein:Creatinine Ratio
Summary of Diabetes Self-Care Activities Scale (SDSCA) | 12 months
  SDSCA is a measure of self-care behaviors in diabetes. It is divided into the following five domains: Diet , Physical Activity, Blood Sugar Testing, Medication Adherence, and Smoking. There are 11 items, with each scored from 0 -7. Higher scores indicate a better outcome. Smoking status is scored using Yes/No.
2-item Diabetes Distress Scale (DDS-2) | 12 months
  The 2-item Diabetes Distress Scale (DDS-2) measures Diabetes Related Distress. It includes two items, each scored from 1 - 6. Higher scores indicate a worse outcome
Diabetes Empowerment Scale (DES-SF) | 12 months
  Diabetes Empowerment Scale (DES-SF) is a measure of diabetes empowerment, consisting of 8 items, each scored from 1 - 5. Higher scores indicate a better outcome.
EuroQol group 5-Dimension 5-Level Scale (EQ-5D-5L) | 12 months
  The EQ-5D-5L is a measure of Health-related quality of life. It is divided into the following five domains: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression (each question scored from 1-5, Higher scores indicate a worse outcome), as well as a Visual Analog Scale (scored from 0- 100, Higher scores indicate a better outcome.)
5 questions from the Patient Satisfaction Questionnaire-III | 3 months
  5 questions from the Patient Satisfaction Questionnaire-III are used as a measure of patient satisfaction in the PACT Arm. It includes five items, each scored between 1-5. Higher scores indicate a worse outcome.
CollaboRATE scale. | 3 months
  The collaboRATE scale is a measure of shared-decision making. It includes three items, each scored between 0-9. Higher scores indicate a better outcome.
Referral to community exercise programs | 12 months
  Patient-reported information for referral to community exercise programs
Adverse events | 12 months
  Patient-reported hypoglycaemic episodes requiring emergency department visit and/or admissions to hospital
Drugs Prescribed | 24 months
  Drug prescribed, dosage, and cost
Costs and resource utilisation | 24 months
  Health-service utilisation costs, training costs, laboratory tests costs, medication costs

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Kay Wye Wong, MBBS, Principal Investigator — National Healthcare Group Polyclinics
Locations (3):
- Singapore (3):
  - NHGP Geylang Polyclinic, Singapore
  - NHGP Ang Mo Kio Polyclinic, Singapore
  - NHGP Woodlands Polyclinic, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ministry of Health S. The White Paper on Healthier SG [Internet]. [cited 2023 Jul 7]. Available from: https://www.healthiersg.gov.sg/resources/white-paper/
- [Background] Ow Yong LM, Koe LWP. War on Diabetes in Singapore: a policy analysis. Health Res Policy Syst. 2021 Feb 8;19(1):15. doi: 10.1186/s12961-021-00678-1. PMID 33557840
- [Background] Ministry of Health S. MOH | National Population Health Survey 2019/20 [Internet]. [cited 2023 Jul 7]. Available from: https://www.moh.gov.sg/resources-statistics/reports/national-survey-2019-20
- [Background] Ministry of Health S. MOH | Singapore Burden of Disease Report 2017 [Internet]. [cited 2023 Jul 7]. Available from: https://www.moh.gov.sg/resources-statistics/singapore-burden-of-disease-report-2017
- [Background] Png ME, Yoong J, Phan TP, Wee HL. Current and future economic burden of diabetes among working-age adults in Asia: conservative estimates for Singapore from 2010-2050. BMC Public Health. 2016 Feb 16;16:153. doi: 10.1186/s12889-016-2827-1. PMID 26880337
- [Background] Ang YG, Yap CW, You AX. Lifetime cost for type 2 diabetes mellitus in Singapore. J Diabetes. 2018 Apr;10(4):296-301. doi: 10.1111/1753-0407.12604. Epub 2017 Sep 29. PMID 28834603
- [Background] Ministry of Health S. MOH | Top 4 Conditions of Polyclinic Attendances [Internet]. [cited 2023 Jul 7]. Available from: https://www.moh.gov.sg/resources-statistics/singapore-health-facts/top-4-conditions-of-polyclinic-attendances
- [Background] Ministry of Health S. MOH CLINICAL PRACTICE GUIDELINES ON DIABETES MELLITUS [Internet]. [cited 2023 Jul 7]. Available from: https://www.moh.gov.sg/hpp/doctors/guidelines/GuidelineDetails/cpgmed_diabetes_mellitus
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] American Diabetes Association. 4. Lifestyle Management: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S38-S50. doi: 10.2337/dc18-S004. PMID 29222375
- [Background] Choi TS, Davidson ZE, Walker KZ, Lee JH, Palermo C. Diabetes education for Chinese adults with type 2 diabetes: A systematic review and meta-analysis of the effect on glycemic control. Diabetes Res Clin Pract. 2016 Jun;116:218-29. doi: 10.1016/j.diabres.2016.04.001. Epub 2016 Apr 26. PMID 27321339
- [Background] Association of Diabetes Care and Education Specialists; Kolb L. An Effective Model of Diabetes Care and Education: The ADCES7 Self-Care Behaviors. Sci Diabetes Self Manag Care. 2021 Feb;47(1):30-53. doi: 10.1177/0145721720978154. PMID 34078208
- [Background] Skovlund SE, Peyrot M, on behalf of the DAWN International Advisory Panel. The Diabetes Attitudes, Wishes, and Needs (DAWN) Program: A New Approach to Improving Outcomes of Diabetes Care. Diabetes Spectr. 2005 Jul 1;18(3):136-42.
- [Background] Wong SKW. Providing care for young adults with type 2 diabetes in primary care settings in Singapore: a multi-faceted study. 2022 [cited 2023 Jul 7]; Available from: https://dr.ntu.edu.sg/handle/10356/163576
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Williams GC, Freedman ZR, Deci EL. Supporting autonomy to motivate patients with diabetes for glucose control. Diabetes Care. 1998 Oct;21(10):1644-51. doi: 10.2337/diacare.21.10.1644. PMID 9773724
- [Background] Silva MN, Vieira PN, Coutinho SR, Minderico CS, Matos MG, Sardinha LB, Teixeira PJ. Using self-determination theory to promote physical activity and weight control: a randomized controlled trial in women. J Behav Med. 2010 Apr;33(2):110-22. doi: 10.1007/s10865-009-9239-y. Epub 2009 Dec 11. PMID 20012179
- [Background] Pillay J, Armstrong MJ, Butalia S, Donovan LE, Sigal RJ, Vandermeer B, Chordiya P, Dhakal S, Hartling L, Nuspl M, Featherstone R, Dryden DM. Behavioral Programs for Type 2 Diabetes Mellitus: A Systematic Review and Network Meta-analysis. Ann Intern Med. 2015 Dec 1;163(11):848-60. doi: 10.7326/M15-1400. Epub 2015 Sep 29. PMID 26414227
- [Background] Huffman MH. Advancing the Practice of Health Coaching: Differentiation From Wellness Coaching. Workplace Health Saf. 2016 Sep;64(9):400-3. doi: 10.1177/2165079916645351. Epub 2016 May 12. PMID 27174131
- [Background] Pirbaglou M, Katz J, Motamed M, Pludwinski S, Walker K, Ritvo P. Personal Health Coaching as a Type 2 Diabetes Mellitus Self-Management Strategy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Health Promot. 2018 Sep;32(7):1613-1626. doi: 10.1177/0890117118758234. Epub 2018 Apr 15. PMID 29658286
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Monica 1776 Main Street Santa, California 90401-3208. Patient Satisfaction Questionnaires (PSQ-III and PSQ-18) [Internet]. [cited 2023 Jul 19]. Available from: https://www.rand.org/health-care/surveys_tools/psq.html
- [Derived] Lee JHB, Yeo LS, Soon WSW, Ding SY, Ge L, Pereira MJ, Foo SCL, Chern CWF, Wong SKW. A cluster randomized trial of a health coach-led patient activation program in type 2 diabetes in Singapore - a study protocol. BMC Prim Care. 2025 Dec 1;26(1):386. doi: 10.1186/s12875-025-03061-z. PMID 41327015
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639